CLINICAL TRIAL: NCT01935505
Title: Study on the Model of Smoking Cessation Intervention and Service Ability Improvement in General Hospital
Brief Title: Study on the Model of Smoking Cessation Intervention and Service Ability Improvement
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yao He, Institute of Geriatrics, Chinese PLA General Hospital
Other Study IDs: IGPLAGH301YaoHe
Record Dates: First submitted 2013-08-25; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; intervention model; Chinese; quitting rate
MeSH Terms: conditions — Smoking Cessation | interventions — Referral and Consultation; Tobacco Use Cessation Devices; Bupropion; Varenicline

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Consulting group: The physicians adopted a non-directive approach, included the five 'A' (ask, advice, assess, assist and arrange), assessing the stage of readiness in quitting smoking, strengthening clients' motivation to quit smoking using the five 'R' (relevance, risks, rewards, roadblocks and repetition) approach, and providing advice to overcome psychological craving, psychological dependence and social-cultural factors associated with tobacco dependency. Each smoker takes more than 30 min to complete the intervention.
  Interventions: Behavioral: Consulting
- Drug intervention group: According to the smokers' level of nicotine dependency, disease history, cigarette consumption, prescription of drugs were provided, Nicotine Replacement Therapy, bupropion and varenicline.
  Interventions: Behavioral: Consulting; Drug: Nicotine patch; Behavioral: Telephone intervention
- Telephone intervention group: Smokers received follow-up by a counselor at 1 week, 1, 3, 6 months and 1, 2 years using a detailed questionnaire by telephone interview. At each follow-up, we collected data, asked whether the smokers have any problem with drug use or other problems, provided problem-oriented suggestions or advice as appropriate, encouraged them to insist.
  Interventions: Behavioral: Consulting; Behavioral: Telephone intervention
- Consulting+Telephone+Drug intervention: All the interventions above are include in this group
  Interventions: Behavioral: Consulting+Telephone+Drug intervention

INTERVENTIONS:
Behavioral: Consulting — The physicians adopted a non-directive approach, included the five 'A' (ask, advice, assess, assist and arrange), assessing the stage of readiness in quitting smoking, strengthening clients' motivation to quit smoking using the five 'R' (relevance, risks, rewards, roadblocks and repetition) approach, and providing advice to overcome psychological craving, psychological dependence and social-cultural factors associated with tobacco dependency. Each smoker takes more than 30 min to complete the intervention.
  Groups: Consulting group; Drug intervention group; Telephone intervention group
Drug: Nicotine patch — According to the smokers' level of nicotine dependency, disease history, cigarette consumption, prescription of drugs were provided, Nicotine Replacement Therapy, bupropion and varenicline.
  Other Names: Nicotine Replacement Therapy: Nicotine patch; bupropion; varenicline
  Groups: Drug intervention group
Behavioral: Telephone intervention — Smokers received follow-up by a counselor at 1 week, 1, 3, 6 months and 1, 2 years using a detailed questionnaire by telephone interview. At each follow-up, we collected data, asked whether the smokers have any problem with drug use or other problems, provided problem-oriented suggestions or advice as appropriate, encouraged them to insist.
  Groups: Drug intervention group; Telephone intervention group
Behavioral: Consulting+Telephone+Drug intervention — Include all the above interventions
  Groups: Consulting+Telephone+Drug intervention

SUMMARY:
This is a observation non-randomized control trial, and a follow-up study on the smoking cessation.

DETAILED DESCRIPTION:
This is a observation non-randomized control trial, and a follow-up study on the smoking cessation.

To study the intervention methods of smoking cessation in a general hospital and to evaluate their effects. Four methods of specialist intervention of smoking cessation clinic, short-time intervention in out patients, free medical intervention and group intervention were adopted for different smokers, with health counseling, psychological intervention and drug treatment. The intervention effect was evaluated by standard methods.

The whole project will last for 10 years in total, from Oct.2008 to Dec.2018. During the running, each quitter received follow-up at 1 week, 1, 3, 6 months and 1, 2 years using a detailed questionnaire by telephone interview, an expected average of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* current smoker aged 18 years or above, Chinese,
* agreed to participate in the follow-up and signed an informed consent form.

Exclusion Criteria:

* cognitively impaired and with severe diseases,
* occasional or daily smoker,
* Disagree and non-signed an informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital-based population
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-10; Primary Completion 2013-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
quitting rate | up to 10 years
  The whole project will last for 10 years in total, from Oct.2008 to Dec.2018. During the running, each participant will be followed by telephone tracking, an expected average of 2 years.

SECONDARY OUTCOMES:
decrease of tobacco consumption | up to 10 years

OTHER OUTCOMES:
changes of Knowledge Attitude and Practice | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yao He, MD, PhD, Principal Investigator — Institute of Geriatrics, Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Jiang B, He Y, Zuo F, Wu L, Liu QH, Zhang L, Zhou CX, Cheng KK, Chan SS, Lam TH. Effectiveness of varenicline and counselling for smoking cessation in an observational cohort study in China. BMJ Open. 2016 Jan 6;6(1):e009381. doi: 10.1136/bmjopen-2015-009381. PMID 26739730